CLINICAL TRIAL: NCT05372796
Title: Effects of Transcutaneous Occipital Nerve Stimulation and Instrument-Assisted Soft Tissue Mobilization in Chronic Migraine
Brief Title: The Effects of Transcutaneous Occipital Nerve Stimulation and Instrument-Assisted Soft Tissue Mobilization on Patients With Chronic Migraine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emine Atıcı (Other)
Collaborators: KTO Karatay University (Other)
Responsible Party: Sponsor-Investigator, Emine Atıcı, Principal Investigator, Okan University
Organization: Okan University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 007
Record Dates: First submitted 2022-04-28; First posted 2022-05-13 (Actual); Last update posted 2022-05-13 (Actual); Status verified 2022-05

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group (Experimental): participants were given home exercise (once a day for 5 weeks)
  Interventions: Other: home exercise
- IASTM (instrument-assisted soft tissue mobilization) (Experimental): IASTM was applied to the patients (M. Sternocleidomastoideus, M. Trapezius, M. Paraspinales and M. Levator Scapula) in the IASTM group twice a week for 5 weeks.
  Interventions: Other: IASTM
- OTES (Occipital Transcutenous Electric Stimulation) (Experimental): Participants in the OTES group were treated with a Chattanooga direct Tens device (DJO UK Ltd, Guildford Surrey, United Kingdom) 3 times a week for 5 weeks. Four self-adhesive 40*40 mm sized electrodes were attached to the occipital region of the patients bilaterally, covering the occipital nerves. The current intensity was adjusted according to the patient. The current intensity started from 0 mA and the current intensity was increased one by one every 30 seconds, the patient was allowed to tolerate the current by giving current without muscle twitching or harmful stimulation. The current frequency was determined as 2/100 Hz. Square waves at 2 Hz were applied for 3 seconds followed by an automatic shift to 100 Hz for another 3 seconds.
  Interventions: Device: Chattanooga direct Tens device (DJO UK Ltd, Guildford Surrey, United Kingdom)

INTERVENTIONS:
Other: IASTM — instrument-assisted soft tissue mobilization
  Arms: IASTM (instrument-assisted soft tissue mobilization)
Other: home exercise — home exercise
  Arms: Control Group
Device: Chattanooga direct Tens device (DJO UK Ltd, Guildford Surrey, United Kingdom) — OTES (Occipital Transcutenous Electric Stimulation)
  Arms: OTES (Occipital Transcutenous Electric Stimulation)

SUMMARY:
In this study, it was aimed to examine the effects of two different treatments applied to the neck region, which have been popular in recent years, on migraine.The study included 45 female patients aged 20-50 years with migraine complaints. The patients were divided into 3 randomized groups: control group (n=15), Instrument-Assisted Soft tissue Mobilization (EDYDM) group (n=15) and on Occipital nerve TENS (OTES) group(n=15).Each group was given home exercise to their treatment. Home exercises applied 1 time per day for 5 weeks. Each exercise in the exercise program was performed with 10 repetitions

ELIGIBILITY:
Inclusion Criteria:

* Be between the ages of 20-50
* International Classification of headache disorders, Third Edition (beta), using the criteria to be diagnosed with migraine without aura,
* migraine with a history of being at least an annual,
* VAS neck pain to be on Level 4,
* the hit-6 score is greater than 56

Exclusion Criteria:

* receiving pharmacological or non-pharmacological treatment regularly in the last three months,
* using a pacemaker,
* being an epileptic or severely psychiatric patient,
* conducting a surgical operation from the neck region,
* cervical disc degeneration or prolapse, the presence of different diagnoses of headaches

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-01-30 (Actual); Study Completion 2022-02-26 (Actual)

PRIMARY OUTCOMES:
Visuel Analog Skale | Change from Baseline Pain at 5 weeks
  VAS is a one-dimensional scale used to determine the severity of pain. The patient is asked to mark the pain he feels on a straight line of 10 cm. the value '0" means that there is no pain at all, and the value "10" means the most severe pain

SECONDARY OUTCOMES:
Headache effect test (HIT-6) | Change from baseline headache at 5 weeks
  The Headache Impact Test-6 (HIT-6) has been developed to measure the factors contributing to headache and provides quantitative information about the impact of headache. HIT-6 consists of 6 items: pain, social functioning, role function, vitality, cognitive function and psychological distress. Scores ranging from 36 to 78 are obtained from the test Dec High scores indicate that the patient's headache negatively affects his daily life
Pittsburgh sleep quality index (PQI) | change from baseline sleep at 5 weeks
  The Pittsburgh sleep quality index (PQI) consists of 24 questions in total. The individual himself answers 19 of these questions. The remaining five questions are answered by the person staying with him, if the person is left alone, they are evaluated for informational purposes and are not added as scoring. There are seven dimensions in the index, namely subjective sleep quality, sleep latency, sleep duration, habitual sleep pattern, sleep disorder status, drug use to fall asleep, daytime dysfunction. The question of each dimension Dec a score between 0 and 3. A total score of 7 dimensions in total gives a sleep quality score. The total score is the range from 0 to 21. The sleep quality of people with a score total below 5 is 'good'; for those with more than 5, their sleep quality is interpreted as 'bad
SF 36 | Change from baseline quality of life at 5 weeks
  The SF-36 quality of life index is a scale that evaluates a person's general health status. 2 basic parameters (mental and physical) and 8 sub-parameter (emotional function, physical function, physical role, social function, mental health, general health, vitality, and pain) to rate on the total consists of 36 questions. From 0 to 100 points can be obtained from each parameter. High scores indicate that a person's quality of life is good

CONTACTS AND LOCATIONS:
Locations (1):
- Emine Atıcı, Tuzla, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No